CLINICAL TRIAL: NCT00057161
Title: Homelessness Prevention: Psychiatric Care With Representative Payeeship
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIR 98-154
Record Dates: First submitted 2003-03-27; First posted 2003-03-28 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-02

CONDITIONS: Mental Illness
MeSH Terms: conditions — Mental Disorders | interventions — Case Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Behavioral: Coordinated Representative Payeeship with Case Management

INTERVENTIONS:
Behavioral: Coordinated Representative Payeeship with Case Management

SUMMARY:
Money management is a neglected issue in maintaining persons with mental illness in the community. This randomized controlled trial (RCT) assessed whether a community-based representative payee program, i.e., money management of Social Security and/or VA benefits, coordinated with VA psychiatric care (CO-RP) could be more effective than customary treatment for veterans who had no representative payee.

DETAILED DESCRIPTION:
Background:

Money management is a neglected issue in maintaining persons with mental illness in the community. This randomized controlled trial (RCT) assessed whether a community-based representative payee program, i.e., money management of Social Security and/or VA benefits, coordinated with VA psychiatric care (CO-RP) could be more effective than customary treatment for veterans who had no representative payee.

Objectives:

After 184 subjects were randomly assigned to CO-RP experimental group or customary care control group, hypotheses were that the CO-RP group would experience: 1) more frequent enrollment in the representative payee program, 2) improved residential status, 3) improved health-related quality of life, including less mental illness symptomatology, 4) less substance abuse, 5) improved money management.

Methods:

Six-month interviews were completed on 152 of 184 possible subjects (83%) and 12-month interviews were completed on 149 of 184 possible subjects (81%). The six and twelve-month outcomes were analyzed with analysis of covariance using data from the baseline pretest.

Status:

Completed.

ELIGIBILITY:
Inclusion Criteria:

Severe mental illness; Inability to manage money; VA patient

Exclusion Criteria:

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Study Completion 2004-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kendon J. Conrad, MA PhD MSPH, Principal Investigator — Edward Hines Jr. VA Hospital, Hines, IL
Locations (1):
- Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois, United States

REFERENCES:
- [Result] Conrad KJ, Lutz G, Matters MD, Donner L, Clark E, Lynch P. Randomized trial of psychiatric care with representative payeeship for persons with serious mental illness. Psychiatr Serv. 2006 Feb;57(2):197-204. doi: 10.1176/appi.ps.57.2.197. PMID 16452696
- [Result] Conrad KJ, Matters MD, Luchins DJ, Hanrahan P, Quasius DL, Lutz G. Development of a Money Mismanagement Measure and cross-validation due to suspected range restriction. J Appl Meas. 2006;7(2):206-24. PMID 16632903
- [Result] Conrad KJ, Wright BD, McKnight P, McFall M, Fontana A, Rosenheck R. Comparing traditional and Rasch analyses of the Mississippi PTSD Scale: revealing limitations of reverse-scored items. J Appl Meas. 2004;5(1):15-30. PMID 14757989